CLINICAL TRIAL: NCT06636565
Title: Comparison of Pulmonary Function, Exercise Capacity, and Physical Activity Level Between Children With Hemophilia and Healthy Controls
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aslihan Cakmak-Onal, Principal Investigator, Hacettepe University
Other Study IDs: FTREK24/65
Record Dates: First submitted 2024-10-07; First posted 2024-10-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2024-10

CONDITIONS: Hemophilia; Healthy Children
Keywords: Hemophilia; Exercise capacity; Pulmonary function
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Hemophilia: Children with hemophilia
  Interventions: Other: No intervention
- Healthy children: Healthy children
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Hemophilia is a rare X-linked congenital bleeding disorder characterized by deficiency of clotting factor VIII (hemophilia A) or deficiency of factor IX (hemophilia B) with complex diagnosis and management. Participation in physical activity is still limited in children with hemophilia, probably due to protective attitudes of families/patients and avoidance of activity, and possibly also as a result of chronic pain. Exercise capacity has been identified as a protective factor against joint problems in hemophilia. Aerobic fitness is associated with better pulmonary function in children. Chronic pain and decreased range of motion due to recurrent bleeding in joints and muscles in hemophilia may indirectly affect posture and respiratory mechanics, leading to impaired pulmonary function. This study aims to compare pulmonary function, exercise capacity, posture, and physical activity level between children with hemophilia and healthy controls and to investigate the relationship between these parameters.

ELIGIBILITY:
Hemophilia group

Inclusion criteria:

* Having been diagnosed with hemophilia and being clinically stable,
* Being between the ages of 8-18,
* Being on prophylaxis treatment (a routine treatment),
* Being 125 cm or taller,
* Being inhibitor negative at the time of enrollment,
* To be able to cooperate with the tests to be performed,
* Being willing to participate in the study.

Exclusion criteria:

* Being inhibitor positive at the time of enrollment,
* Having a history of acute joint bleeding,
* Being unable to bear weight on the extremities,
* Having a history of acute intramuscular bleeding,
* Having undergone radionuclide synovectomy,
* Having a history of surgery on any of the lower extremity joints,
* Having a severe cardiovascular, orthopedic or neurological problem that may affect the assessments.

Control group

Inclusion criteria:

* Not having any known internal or chronic disease
* Being male between the ages of 8-18
* Having full range of motion in the upper extremity
* Having full range of motion in the lower extremity
* Not having any history of injury or surgery in the lower extremity
* Being 125 cm or taller
* Being willing to participate in the study

Exclusion criteria:

* Having any problem that may affect the tests
* Not having full range of motion in the upper extremity
* Having a history of injury or surgery in any of the lower extremity joints
* Having a neurological deficit
* Having pain or movement limitation in the lower extremity

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children with hemophilia and their healthy peers
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2024-07-25 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Forced vital capacity | 1st day
  Pulmonary function test using a spirometer will be performed. Forced vital capacity will be recorded.
Forced expiratory volume in one second | 1st day
  Pulmonary function test using a spirometer will be performed. Forced expiratory volume in one second will be recorded.
Forced expiratory volume in one second/forced vital capacity ratio | 1st day
  Pulmonary function test using a spirometer will be performed. Forced expiratory volume in one second/forced vital capacity ratio will be recorded.
Peak expiratory flow | 1st day
  Pulmonary function test using a spirometer will be performed. Peak expiratory flow will be recorded. will be recorded.
Forced mid-expiratory flow (FEF25-75) | 1st day
  Pulmonary function test using a spirometer will be performed. Forced mid-expiratory flow (FEF25-75) will be recorded. will be recorded.
Hemophilia Joint Health Score | 1st day
  Hemophilia Joint Health Score is a scoring used by physiotherapists in hemophilia treatment centers to detect early hemophilic arthropathy symptoms and to monitor joint health. HJHS consists of edema (0-3), duration of edema (0-1), muscle atrophy (0-2), crepitus during movement (0-2), loss of flexion (0-3), loss of extension (0-3), joint pain (0-2) and evaluation of muscle strength of knees, ankles and elbows (0-4) and global gait score (0-4). The maximum score is 124, with higher scores indicating worse joint health.
Corbin Posture Rating Scale | 1st day
  Corbin Posture Rating Scale and observational posture analysis. It is an assessment consisting of lateral and posterior posture analysis. '0' is excellent, 12 and above indicates poor posture.
Exercise capacity | 1st day
  To assess exercise capacity, a symptom-limited cardiopulmonary exercise test will be performed on a bicycle ergometer using Godfrey protocol. Cardiopulmonary responses and effort perceptions will be recorded. In Godfrey protocol, workload increases are adjusted according to height: workload is increased by 10 W/min for < 125 cm, by 15 W/min for 125-150 cm and by 20 W/min for >150 cm.
Physical activity level | 1st day
  The Physical Activity Questionnaire for Children (PAQ-C) and the Physical Activity Questionnaire for Adolescents (PAQ-A) will be used to assess physical activity levels. The Turkish versions of these assessment tools have been shown to be valid and reliable.

CONTACTS AND LOCATIONS:
Overall Officials: Aslihan Cakmak-Onal, PhD, PT, Principal Investigator — Hacettepe University; Ebru Calik-Kutukcu, PhD, PT, Study Director — Hacettepe University; Hande Guney-Deniz, PhD, PT, Study Chair — Hacettepe University; Ş. Selin Aytac-Eyupoglu, MD, Study Chair — Hacettepe University; Firat Tan, MSc, PT, Principal Investigator — Ataturk University
Locations (1):
- Hacettepe University Faculty of Physical Therapy and Rehabilitation, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No